CLINICAL TRIAL: NCT05607251
Title: Salivary Alkaline Phosphatase as a Biomarker for Dental Caries in A Group of Egyptian Children With Different Growth Rates: A Descriptive Cross-Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Ahmed Abdelrahman, General Dentist, Cairo University
Other Study IDs: CUP1/11/2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There is no intervention as this is an observational study

SUMMARY:
Aim of the study:

1. Assess the correlation between salivary alkaline phosphatase levels and dental caries.
2. Assess the effect of growth of children on the levels of salivary alkaline phosphatase enzyme.
3. Assess the effect of growth of children on caries experience and severity.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 8 years old.
* Children with and without previous dental visits.

Exclusion Criteria:

* Children with any systemic or mental illness.
* Children whose parents refuse to sign the informed consent.
* Children who will not cooperate on participation

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged between 6-8 years.
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Salivary Alkaline Phosphatase levels in children with and without dental caries | 2 months
  Measured by spectrophotometry (unit: U/L)

SECONDARY OUTCOMES:
Caries index | 2 months
  Measured by DMFT and deft (unit: scores)
Caries severity | 2 months
  Measured by ICDAS (unit: scores)

IPD SHARING:
Plan to Share IPD: Undecided